CLINICAL TRIAL: NCT06341114
Title: A Multicenter, Open-label Phase Ib-II Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy of the Combination of BAT8008 With BAT1308 in Patients With Advanced Solid Tumors
Brief Title: A Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy of the Combination of BAT8008 With BAT1308 in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAT-8008-1308-001-CR
Record Dates: First submitted 2024-03-14; First posted 2024-04-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- A/ Standard 3+3 2.1mg/kg of BAT8008 (Experimental): Drug: BAT8008， Dosage: 2.1mg/kg, Frequency: once every 2 weeks, Duration: 1year
  Interventions: Drug: BAT8008 injection
- B/ Standard 3+3 2.4mg/kg of BAT8008 (Experimental): Drug: BAT8008， Dosage: 2.4mg/kg, Frequency: once every 2 weeks, Duration: 1year
  Interventions: Drug: BAT8008 injection
- Standard 3+3 200mg of BAT1308 (Experimental): Drug: BAT1308， Dosage: 200mg, Frequency: once every 2 weeks, Duration: 1year
  Interventions: Drug: BAT1308 injection
- A/ Standard 3+3 1.8mg/kg of BAT8008 (Experimental): Drug: BAT8008， Dosage: 1.8mg/kg, Frequency: Day1 and Day8，once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8008 injection
- B/ Standard 3+3 2.1mg/kg of BAT8008 (Experimental): Drug: BAT8008， Dosage: 2.1mg/kg, Frequency: Day1 and Day8，once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8008 injection
- Standard 3+3 300mg of BAT1308 (Experimental): Drug: BAT1308， Dosage: 300mg Frequency: Day1 and Day8，once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT1308 injection

INTERVENTIONS:
Drug: BAT8008 injection — BAT8008 for injection is a sterile, preservative-free lyophilized powder packaged in vials, with each vial containing 100 mg,Prior to infusion, reconstitute with 5 milliliters of sterile water for injection. After reconstitution, a clear to slightly opalescent, colorless to pale yellow solution with a final concentration of 20 mg/mL can be obtained.
  Arms: A/ Standard 3+3 1.8mg/kg of BAT8008; A/ Standard 3+3 2.1mg/kg of BAT8008; B/ Standard 3+3 2.1mg/kg of BAT8008; B/ Standard 3+3 2.4mg/kg of BAT8008
Drug: BAT1308 injection — One vial of 4 mL of concentrate contains 100 mg of BAT1308.
  Arms: Standard 3+3 200mg of BAT1308; Standard 3+3 300mg of BAT1308

SUMMARY:
The study, led by Zhejiang Cancer Hospital and sponsored by Bio-Thera Solutions, Ltd., is an exploratory multicenter, open-label phase Ib-II clinical trial evaluating the safety, tolerability, pharmacokinetic characteristics, and preliminary efficacy of the combination of BAT8008 with BAT1308 in patients with advanced solid tumors.

This study aims to explore the safety, tolerability, and pharmacokinetic characteristics of BAT8008 combined with BAT1308 in patients with advanced solid tumors, determine the maximum tolerated dose (MTD), provide recommended doses and reasonable dosing regimens for subsequent clinical studies, and preliminarily evaluate the antitumor efficacy.

The study is divided into two stages. The first stage will use a "3+3" dose escalation design to explore the safety and tolerability of the investigational drugs. In the second stage, based on the preliminary safety and efficacy results from the first stage, appropriate doses and tumor types will be selected for expansion studies within the safety dose range to further investigate the safety and clinical efficacy of BAT8008+BAT1308 and provide evidence for subsequent clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender not specified;
2. Voluntary signing of the informed consent form;
3. Must be pathologically diagnosed by histology or cytology, with standard treatment failure or absence of standard treatment, intolerance to standard treatment, or refusal of standard treatment for advanced or metastatic epithelial solid tumor patients. Expanded Research Phase: Divided into two cohorts (the sponsor may expand or delete cohorts of tumor types based on real-time study results): Cohort A: Locally advanced or metastatic triple-negative breast cancer diagnosed by histology or cytology, and subjects who cannot be cured by radical resection or radiotherapy, and have used at least one systemic chemotherapy regimen for advanced or metastatic disease. Cohort B: Other advanced or metastatic epithelial solid tumor patients who are intolerant or refuse standard treatment, prioritizing the following types: non-squamous non-small cell lung cancer, gastric adenocarcinoma, esophageal cancer, small cell lung cancer, cervical cancer, and head and neck squamous cell carcinoma.
4. According to RECIST 1.1 criteria, there must be evaluable tumor lesions in the dose escalation phase, and at least one measurable tumor lesion in the dose expansion phase;
5. Eastern Cooperative Oncology Group (ECOG) performance status score required is 0 or 1;
6. Investigator-assessed expected survival period ≥ 12 weeks;
7. Must have sufficient organ and bone marrow reserve function, defined as follows:

   Hematology (no blood transfusions, hematopoietic growth factors, or drugs to correct blood cell counts within 14 days prior to first dose):

   Absolute neutrophil count (ANC) ≥ 1.5 × 10^9 /L Platelet count ≥ 90 × 10^9 /L Hemoglobin ≥ 90 g/L

   Coagulation:

   International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5×ULN (for patients not receiving anticoagulation therapy) Patients receiving oral anticoagulant therapy with an INR of 2~3 can be included

   Liver function:

   Total bilirubin (TBIL) ≤ 1.5×ULN For liver cancer or liver metastases, ≤2×ULN Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN For liver cancer or liver metastases, ≤5×ULN

   Renal function:

   Serum creatinine ≤ 1.5×ULN or estimated glomerular filtration rate > 50 ml/min (using Cockcroft-Gault or modified MDRD formula, see appendix) Urine protein: Urinalysis suggests urine protein < 2+ or urine protein quantification < 1g
8. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose and be willing to use effective contraception methods during the study period until 6 months after the last dose; male patients must agree to use effective contraception methods during the study period until 6 months after the last dose; postmenopausal women must have been amenorrheic for at least 12 months to be considered not of childbearing potential;
9. Willing to provide past archived or fresh tumor tissue samples (if there is no archived tumor tissue in the past, and the investigator assesses that there is a significant risk in obtaining fresh or metastatic tumor tissue specimens, exemption may be granted). Immunohistochemical confirmation of PDL1 and Trop2 expression levels is not required before enrollment, but the sponsor requires the collection of biopsy or archived tumor tissue samples to determine PDL1 and Trop2 expression levels;
10. Able to understand the requirements of the trial, willing, and able to comply with the trial and follow-up arrangements.

Exclusion Criteria：

1. Within the first 4 weeks prior to the initial administration of the investigational drug, having received experimental drug therapy or participated in clinical studies of medical devices.
2. Within the first 4 weeks prior to the initial administration of the drug, having undergone chemotherapy, curative radiotherapy (palliative radiotherapy should be completed within 2 weeks prior to the initial drug administration), biological therapy, endocrine therapy, immunotherapy, or other anti-tumor treatments; 2) For fluoropyrimidine drugs and small molecule targeted drugs, within 2 weeks prior to the initial administration of the investigational drug or within 5 half-lives of the drug (whichever is longer); 3) Within 42 days prior to the initial administration of the investigational drug for nitrosourea drugs or mitomycin C.
3. Having received, within 1 week prior to drug administration, traditional Chinese medicine or treatment explicitly indicated in the drug instructions approved by the NMPA for its anti-tumor functions, or having a clear record in medical history of herbal treatment for anti-tumor purposes.
4. Prior anti-tumor therapy resulting in adverse events (AEs) (CTCAE 5.0) still at > Grade 1 before the initial administration of the investigational drug, excluding toxicities judged by the investigator to pose no safety risk, such as alopecia, Grade 2 peripheral neuropathy, etc.
5. Needing major surgery within the first 4 weeks prior to the initial administration of the investigational drug (excluding procedures for diagnosis) or anticipated major surgery during the study period.
6. Patients who have previously received Trop2-ADC with small molecule toxins that are topoisomerase I inhibitors.
7. Having experienced ≥ Grade 3 immune-related adverse events (irAEs) in the past or having discontinued immunotherapy due to irAEs of any grade.
8. Individuals with a history of allogeneic cell or solid organ transplantation.
9. Patients with primary central nervous system tumors or symptomatic central nervous system metastases, a history of or currently present meningeal metastases, or a history of seizures. If brain metastases are stable after treatment and there are no new lesions at least 4 weeks before medication, or if asymptomatic lesions are detected for the first time within 4 weeks and the investigator determines disease stability, or if the investigator decides to discontinue corticosteroid treatment 7 days before the initial administration of the investigational drug, then it is allowed.
10. Any other active malignant tumors within 5 years before the initial administration of the drug, except for locally cured tumors (such as basal cell carcinoma, squamous cell carcinoma of the skin, superficial bladder cancer, or ductal carcinoma in situ of the breast).
11. Occurrence of the following cardiovascular diseases within 6 months before the initial administration of the drug: symptomatic heart failure of New York Heart Association (NYHA) class 2 or higher, left ventricular ejection fraction (LVEF) <50%, unstable arrhythmias or unstable angina, myocardial infarction requiring treatment, pulmonary embolism, uncontrolled hypertension (defined in this protocol as systolic blood pressure >160mmHg and/or diastolic blood pressure >100mmHg despite optimal antihypertensive therapy, and assessed by the investigator to have clinical significance), QTcF >480ms on 12-lead electrocardiogram (QTcF calculated using the Fridericia correction formula).
12. Presence of any other severe underlying diseases (e.g., Gilbert's syndrome, poorly controlled diabetes, active peptic ulcer, unstable controlled seizures, cerebrovascular events/gastrointestinal bleeding within 3 months before the initial administration of the drug, coagulation disorders with severe symptoms or signs), as judged by the investigator to potentially affect the subject's participation in the study, treatment, and follow-up, affect subject compliance, or potentially lead to occurrences of drug-related complications in the subjects.
13. History of non-infectious pneumonia/pulmonary inflammation requiring glucocorticoid treatment, current interstitial lung disease (ILD), or subjects in the screening period with suspected ILD/pulmonary inflammation that cannot be ruled out by imaging examinations.
14. Patients with a history of autoimmune diseases (except for autoimmune thyroid diseases and type I diabetes that can be treated with hormone replacement therapy).
15. Received systemic corticosteroids (prednisone > 10mg/day or equivalent) or other immunosuppressive agents within 14 days prior to the initial use of the investigational drug; exceptions include the following: use of topical, ocular, intra-articular, intranasal, or inhaled corticosteroids, short-term prophylactic use of corticosteroids (duration not exceeding 2 weeks, e.g., for contrast allergy prophylaxis).
16. Untreated or actively treated tuberculosis subjects, including but not limited to pulmonary tuberculosis; subjects who have undergone standard anti-tuberculosis treatment and have been confirmed by the investigator to be cured may be included.
17. Experienced severe infection within 4 weeks prior to the initial administration of the drug or active infection within 2 weeks.
18. Subjects with the following infectious diseases: Human Immunodeficiency Virus (HIV) infection; active Hepatitis B Virus infection [Hepatitis B Surface Antigen (HBsAg) positive, with Hepatitis B Virus Deoxyribonucleic Acid (HBV-DNA) > 200 IU/ml or 10^3 copies/ml or within the upper limit of normal value determined by the study center]; Hepatitis C Virus infection [HCV antibody and Hepatitis C Virus Ribonucleic Acid (HCV-RNA) positive]; positive syphilis treponemal antibody and RPR/TRUST positive.
19. Newly diagnosed thromboembolic events requiring treatment within 6 months (patients with stable lower extremity deep vein thrombosis or port-related thrombosis are allowed to be included).
20. Difficult-to-control pleural effusion, pericardial effusion, or ascites requiring repeated drainage surgery (monthly or more frequently).
21. Known hypersensitivity reaction or delayed allergic reaction to any component of the investigational drug.
22. Known occurrence of ≥ Grade 3 allergic reactions to macromolecular protein preparations/monoclonal antibodies.
23. History of mental illness, substance abuse, alcoholism, or drug abuse that may affect trial results.
24. Pregnant or lactating women or individuals planning to conceive.
25. Other conditions deemed inappropriate for participation in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-04-03 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | The first administration cycle(21 days)
  DLT events and their incidence.
vital signs | Through study completion, 1 year
  Number of participants with abnormal vital signs
Physical examination | Through study completion, 1 year
  Number of participants with abnormal physical examination
Adverse events | From the first receipt of the investigational drug until 28 (+7) days after the last receipt of the investigational drug or the initiation of a new antitumor therapy, whichever occurs earlier，assessed up to 1 year
  Number of cases with all adverse medical events that occur after the subject receives the investigational drug assessed by CTCAE V5.0
Clinical laboratory tests | Through study completion, 1 year
  Number of participants with abnormal clinical laboratory tests
Clinical auxiliary tests | Through study completion, 1 year
  Number of participants with abnormal clinical auxiliary tests
Objective response rate (ORR) | Through study completion, 1 year
  Refer to the proportion of subjects defined as complete remission (CR) and partial remission (PR)
Duration of Response(DOR) | Through study completion, 1 year
  DoR is defined as the time between the first assessment of objective remission of a tumor and death from any cause before the first assessment of Disease progression (PD) , reflecting the duration of ORR.
Disease Control Rate (DCR) | Through study completion, 1 year
  The proportion of patients with tumor reduction or stability maintained for a certain period, including cases of complete response (CR), partial response (PR), and stable disease (SD).
Progression Free Survival(PFS) | Through study completion, 1 year
  Progression Free Survival（PFS ）in patients with advanced or recurrent dMMR endometrial cancer treated with BAT1308 combined with platinum-containing chemotherapy were compared with platinum-containing chemotherapy in first-line treatment by IRC according to RECIST V1.1.
Overall Survival(OS) | Through study completion, 1 year
  The time from the date of first administration to the occurrence of death due to any cause. Subjects who were still alive at the time of analysis will use the date of their last contact as the deadline.

SECONDARY OUTCOMES:
Pharmacokinetic | At the end of Cycle 1 Day 1 (C1D1), Cycle 2 Day 1 (C2D1), Cycle 3 Day 1 (C3D1), Cycle 3 Day 2 (C3D2), Cycle 3 Day 3 (C3D3), Cycle 3 Day 8 (C3D8), Cycle 4 Day 1 (C4D1), after Cycle4, Every 4 cycle until 26 cycles (one cycle equals 2 weeks).
  Level of Tmax
Pharmacokinetic | At the end of Cycle 1 Day 1 (C1D1), Cycle 2 Day 1 (C2D1), Cycle 3 Day 1 (C3D1), Cycle 3 Day 2 (C3D2), Cycle 3 Day 3 (C3D3), Cycle 3 Day 8 (C3D8), Cycle 4 Day 1 (C4D1), after Cycle4, Every 4 cycle until 26 cycles (one cycle equals 2 weeks).
  Level of CL
Pharmacokinetic | At the end of Cycle 1 Day 1 (C1D1), Cycle 2 Day 1 (C2D1), Cycle 3 Day 1 (C3D1), Cycle 3 Day 2 (C3D2), Cycle 3 Day 3 (C3D3), Cycle 3 Day 8 (C3D8), Cycle 4 Day 1 (C4D1), after Cycle4, Every 4 cycle until 26 cycles (one cycle equals 2 weeks).
  Level of T1/2
Pharmacokinetic | At the end of Cycle 1 Day 1 (C1D1), Cycle 2 Day 1 (C2D1), Cycle 3 Day 1 (C3D1), Cycle 3 Day 2 (C3D2), Cycle 3 Day 3 (C3D3), Cycle 3 Day 8 (C3D8), Cycle 4 Day 1 (C4D1), after Cycle4, Every 4 cycle until 26 cycles (one cycle equals 2 weeks).
  Level of Cmax
Pharmacokinetic | At the end of Cycle 1 Day 1 (C1D1), Cycle 2 Day 1 (C2D1), Cycle 3 Day 1 (C3D1), Cycle 3 Day 2 (C3D2), Cycle 3 Day 3 (C3D3), Cycle 3 Day 8 (C3D8), Cycle 4 Day 1 (C4D1), after Cycle4, Every 4 cycle until 26 cycles (one cycle equals 2 weeks).
  Level of ADA
Pharmacokinetic | At the end of Cycle 1 Day 1 (C1D1), Cycle 2 Day 1 (C2D1), Cycle 3 Day 1 (C3D1), Cycle 3 Day 2 (C3D2), Cycle 3 Day 3 (C3D3), Cycle 3 Day 8 (C3D8), Cycle 4 Day 1 (C4D1), after Cycle4, Every 4 cycle until 26 cycles (one cycle equals 2 weeks).
  Level of Nab

CONTACTS AND LOCATIONS:
Locations (1):
- Song ZhengBo, Hangzhou, Zhejiang, China